CLINICAL TRIAL: NCT04371614
Title: PTSC: Improving Hypertension Control Among Poor Midlife African American Women
Acronym: PTSC-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: American Institutes for Research (Other); The Gaston & Porter Health Improvement Center, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MD010462 (NIH)
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2020-04

CONDITIONS: Uncontrolled Hypertension; BMI; Stress; Medication Adherence
Keywords: Hypertension; African American women; Lifestyle Modification
MeSH Terms: conditions — Medication Adherence; Hypertension

STUDY DESIGN:
Intervention Model Description: The women are randomly assigned to receive the PTSC intervention or usual care from the FQHC. The intervention last for 3 months. The women are followed for 1 year after receiving the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prime Time Sister Circle Intervention (Active Comparator): The women in this arm participate in a Prime Time Sister Circle (PTSC). The PTSC is a multi-faceted, facilitated, curriculum- and community-based, intensive, support group intervention with 25-30 mid-life African American women per group. PTSC addresses three key modifiable health risk factors for chronic disease: unmanaged stress, physical inactivity, and unhealthy nutritional choices. It also addresses additional risk factors that contribute to unhealthy lifestyles: lack of knowledge or misinformation about major illnesses-cardiovascular disease (CVD), hypertension, diabetes, cancer, stress and depression-and the failure of African American women to prioritize their health and take proactive steps to manage their health and health outcomes. PTSC gives African American women the information, motivation, tools, skills, and consultative support they need to improve and maintain their health.
  Interventions: Behavioral: Prime Time Sister Circle
- Usual Care (No Intervention): The women in the arm do not receive the intervention but provide data at baseline, 3 months, 9 months and 15 months.

INTERVENTIONS:
Behavioral: Prime Time Sister Circle — The PTSC is a multi-faceted, facilitated, curriculum- and community-based, intensive, support group intervention with 25-30 mid-life African American women per group.
  Arms: Prime Time Sister Circle Intervention

SUMMARY:
African American women are more likely to suffer higher rates of uncontrolled hypertension than non-Hispanic white women. Prime Time Sister Circles® (PTSC) empowers women to proactively manage their blood pressure by promoting the effective use of preventive health care; encouraging self monitoring of blood pressure, and teaching strategies for managing stress, increasing physical activity, and improving nutrition. The 12-week community-based, holistic lifestyle intervention aims to improve blood pressure control by improving health knowledge, health efficacy, and health behaviors. PTSC potentially reduces health care costs through prevention, earlier detection, and improved management of hypertension through a culturally tailored program addressing specific barriers experienced by midlife and late life African American women.

This 5-year study is a collaboration between The Johns Hopkins Center for Health Disparities Solutions (HCHDS), The Gaston & Porter Health Improvement Center, Inc. (GPHIC), and the American Institutes for Research (AIR). The investigators seek to determine the impact and cost-effectiveness of the PTSC intervention among low-income African American women with uncontrolled hypertension. To do this, the investigators will randomly assign 600 women between the ages of 40 and 75 who receive their care from an federally qualified health center (FQHC) to either PTSC (n=300) or a comparison group (n=300) who will receive the PTSC intervention after they have been observed for 15 month. Using data from in person surveys and clinical measures conducted during in-person data collection meetings, the investigative team will determine if PTSC help low-income African American women effectively manage their blood pressure.

DETAILED DESCRIPTION:
African American women suffer significantly higher rates of hypertension than non-Hispanic white women. Forty-six to fifty percent of African American women have hypertension, compared with 31 percent of White women making it a major contributor to disparities in cardiovascular morbidity and mortality in this population from higher rates of complications, i.e., ischemic heart disease, stroke, and end-stage renal disease. Despite these statistics, African American women are less often aware of their diagnosis, less likely to have their blood pressure controlled, and less likely to be treated. From a societal perspective, high blood pressure was estimated to cost the United States approximately $93.5 billion in health care services, medications, and missed work days in 2010.

Public and private health plans, employers, and health care providers are seeking cost-effective approaches to preventing and improving management of uncontrolled hypertension (140/90 and above). Prime Time Sister Circles® (PTSC) empowers women to proactively manage their health by promoting the effective use of preventive health care; providing screening and monitoring of blood pressure and weight, and teaching strategies for managing stress, increasing physical activity, and improving nutrition. The 13-week community-based, holistic lifestyle intervention aims to improve blood pressure control and reduce health care costs through prevention, earlier detection, and improved management of hypertension through a culturally tailored program addressing specific risk factors and barriers experienced by mid to late life African American women.

The primary objective of this research project is to determine the impact and cost-effectiveness of the PTSC intervention among low-income African American women with uncontrolled hypertension. This 5-year study is a collaboration between The Johns Hopkins Center for Health Disparities Solutions (HCHDS), The Gaston & Porter Health Improvement Center, Inc. (GPHIC), and the American Institutes for Research (AIR). Study participants will be recruited from FQHCs in Washington, DC and Baltimore, MD. These FQHCs were chosen because they are medical homes to a large number of low income midlife African American women who have hypertension. The sample, 480 African American women between the ages of 40 and 75 who receive their primary care from a FQHC, will be randomly assigned to receive the PTSC intervention (n=240) or usual care for a FQHC (n=240). Data on blood pressure, health status, health behaviors, and health care utilization will be collected through participant surveys and administrative records from the FQHCs. Blood pressure measurements and surveys will be collected at baseline, 13 weeks (end of program), 9 months (6 months after the end of the program), and 15 months (a year after the end of the program). Administrative records to track health services use and costs will be collected on an ongoing basis over the same time period. These data will be used to address the following specific aims:

Aim 1. Estimate the effectiveness of PTSC compared with usual care on blood pressure control among hypertensive, low-income, mid-to-late life African American women.

Hypothesis 1.1 Patients randomized to PTSC will have better controlled blood pressure than patients who receive usual care at the end of the intervention (13 weeks) and up to one year post intervention (15 months).

Aim 2. Estimate the effectiveness of PTSC on health knowledge, health self-efficacy, and health behaviors that contribute to risks associated with hypertension.

Hypothesis 2.1 Patients randomized to PTSC will demonstrate a greater increase in knowledge of the causes and consequences of high blood pressure than patients receiving usual care.

Hypothesis 2.2 Patients randomized to PTSC will demonstrate a greater increase in health-related self-efficacy than patients receiving usual care.

Hypothesis 2.3 Patients randomized to PTSC will practice more adaptive stress management techniques, increase their level of physical activity, and improve their diets more than patients receiving usual care.

Hypothesis 2.4 Patients randomized to PTSC will monitor their own blood pressure more regularly than patients receiving usual care.

Hypothesis 2.5: Patients randomized to PTSC will be more compliant with taking prescribed hypertension medications than patients receiving usual care.

Aim 3. Test whether there is a cost offset of PTSC for society. Hypothesis 3.1 Patients randomized to PTSC will have fewer unnecessary hospitalizations and emergency rooms visits for cardiovascular related problems than patients receiving usual care.

Hypothesis 3.2 Patients randomized to PTSC will have fewer hospital admissions for cardiovascular related problems than patients receiving usual care.

Hypothesis 3.3 The costs of providing PTSC will be offset by reductions in healthcare costs associated with health improvements for patients randomized to PTSC compared to patients receiving usual care.

FQHCs and other safety net providers are challenged to effectively manage the hypertension of their midlife African American female patients. PTSC may be a viable low-cost, community-based intervention that physicians can use as a resource for their patients to support necessary lifestyle changes and improve their health.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with hypertension (401)
* had a visit to the FQHC within the prior 24 months
* had an elevated blood pressure (140/90 or above) at their last visit
* able to speak English

Exclusion Criteria:

* diagnosed with psychotic disorders (295.42, 295.90)
* diagnosed with dementia (290)
* diagnosed with other nutritional deficiencies (269.9)
* diagnosed with congestive heart failure (428)
* diagnosed with blindness (369.3)

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participate must self identify as female.
Enrollment: 359 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Baseline
  Systolic and Diastolic Blood Pressure
Blood Pressure | 3 months
  Systolic and Diastolic Blood Pressure
Blood Pressure | 9 months
  Systolic and Diastolic Blood Pressure
Blood Pressure | 15 months
  Systolic and Diastolic Blood Pressure
Body Mass Index | Baseline
  Calculation based on height and weight
Body Mass Index | 3 months
  Calculation based on height and weight
Body Mass Index | 9 months
  Calculation based on height and weight
Body Mass Index | 15 months
  Calculation based on height and weight
Waist Circumference | Baseline
  Measured in centimeters
Waist Circumference | 3 months
  Measured in centimeters
Waist Circumference | 9 months
  Measured in centimeters
Waist Circumference | 15 months
  Measured in centimeters

SECONDARY OUTCOMES:
Stress | Baseline
  Perceived Stress Scale Respondents are asked to rate their current stress level on a scale from 1 to 7, where 1 means "not at all stressed," and 7 means "extremely stressed,"
Stress | 3 months
  Perceived Stress Scale Respondents are asked to rate their current stress level on a scale from 1 to 7, where 1 means "not at all stressed," and 7 means "extremely stressed,"
Stress | 9 months
  Perceived Stress Scale Respondents are asked to rate their current stress level on a scale from 1 to 7, where 1 means "not at all stressed," and 7 means "extremely stressed,"
Stress | 15 months
  Perceived Stress Scale Respondents are asked to rate their current stress level on a scale from 1 to 7, where 1 means "not at all stressed," and 7 means "extremely stressed,"
Medication Adherence | Baseline
  Hill-Bone High Blood Pressure Compliance Scale
  This is a scale based on 14 questions where respondents answer
  1. Not at all
  2. Some of the time
  3. Most of the time
  4. All of the time
  The items are additive. The minimum score is 14 indicating most compliance and the maximum is 56 indicating least compliance.
Medication Adherence | 3 months
  Hill-Bone High Blood Pressure Compliance Scale
  This is a scale based on 14 questions where respondents answer
  1. Not at all
  2. Some of the time
  3. Most of the time
  4. All of the time
  The items are additive. The minimum score is 14 indicating most compliance and the maximum is 56 indicating least compliance.
Medication Adherence | 9 months
  Hill-Bone High Blood Pressure Compliance Scale
  This is a scale based on 14 questions where respondents answer
  1. Not at all
  2. Some of the time
  3. Most of the time
  4. All of the time
  The items are additive. The minimum score is 14 indicating most compliance and the maximum is 56 indicating least compliance.
Medication Adherence | 15 months
  Hill-Bone High Blood Pressure Compliance Scale
  This is a scale based on 14 questions where respondents answer
  1. Not at all
  2. Some of the time
  3. Most of the time
  4. All of the time
  The items are additive. The minimum score is 14 indicating most compliance and the maximum is 56 indicating least compliance.
Hypertension Knowledge | Baseline
  COUNSELING AFRICAN AMERICANS TO CONTROL HYPERTENSION (CAATCH)
  This is a 17 item scale where respondents answer True or False to questions about hypertension. The scale has a minimum value of 0 which indicates the respondent is not very knowledgeable about hypertension to 17 which indicates the respondent is very knowledgeable about hypertension.
Hypertension Knowledge | 3 months
  COUNSELING AFRICAN AMERICANS TO CONTROL HYPERTENSION (CAATCH)
  This is a 17 item scale where respondents answer True or False to questions about hypertension. The scale has a minimum value of 0 which indicates the respondent is not very knowledgeable about hypertension to 17 which indicates the respondent is very knowledgeable about hypertension.
Hypertension Knowledge | 9 months
  COUNSELING AFRICAN AMERICANS TO CONTROL HYPERTENSION (CAATCH)
  This is a 17 item scale where respondents answer True or False to questions about hypertension. The scale has a minimum value of 0 which indicates the respondent is not very knowledgeable about hypertension to 17 which indicates the respondent is very knowledgeable about hypertension.
Hypertension Knowledge | 15 months
  COUNSELING AFRICAN AMERICANS TO CONTROL HYPERTENSION (CAATCH)
  This is a 17 item scale where respondents answer True or False to questions about hypertension. The scale has a minimum value of 0 which indicates the respondent is not very knowledgeable about hypertension to 17 which indicates the respondent is very knowledgeable about hypertension.
Functional Status | Baseline
  EuroQol 5
  This is a 5 item scale where respondent are asked whether have problems along five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondent rate each item based on five point scale: (1) no, (2) slight, (3) some, (4) moderate, or (5) extreme. The scale is scored based on a country and population specific valuation that is proprietary. Each dimension make up a digit in a five digit code: 1,1,1,1,1 indicate most healthy state while 5,5,5,5,5 indicates the most unhealthy state.
Functional Status | 15 months
  EuroQol 5
  This is a 5 item scale where respondent are asked whether have problems along five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondent rate each item based on five point scale: (1) no, (2) slight, (3) some, (4) moderate, or (5) extreme. The scale is scored based on a country and population specific valuation that is proprietary. Each dimension make up a digit in a five digit code: 1,1,1,1,1 indicate most healthy state while 5,5,5,5,5 indicates the most unhealthy state.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell J Gaskin, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Baltimore Medical System, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zare H, Ibe CA, Yang M, Porter G, Gaston M, Jones N, Jones W, Rose V, Balamani M, Woods DL, Gaskin DJ. Evaluating the Impact of the Prime Time Sister Circles(R) Intervention on Reducing Depressive Symptoms Among African American Women with Uncontrolled Hypertension. J Gen Intern Med. 2023 Oct;38(13):2879-2887. doi: 10.1007/s11606-023-08288-z. Epub 2023 Jul 27. PMID 37500950
- [Derived] Ibe CA, Haywood DR, Creighton C, Cao Y, Gabriel A, Zare H, Jones W, Yang M, Balamani M, Gaston M, Porter G, Woods DL, Gaskin DJ. Study protocol of a randomized controlled trial evaluating the Prime Time Sister Circles (PTSC) program's impact on hypertension among midlife African American women. BMC Public Health. 2021 Mar 29;21(1):610. doi: 10.1186/s12889-021-10459-8. PMID 33781228
- [Derived] Gabriel A, Zare H, Jones W, Yang M, Ibe CA, Cao Y, Balamani M, Gaston M, Porter G, Woods DL, Gaskin DJ. Evaluating Depressive Symptoms Among Low-Socioeconomic-Status African American Women Aged 40 to 75 Years With Uncontrolled Hypertension: A Secondary Analysis of a Randomized Clinical Trial. JAMA Psychiatry. 2021 Apr 1;78(4):426-432. doi: 10.1001/jamapsychiatry.2020.4622. PMID 33566072